CLINICAL TRIAL: NCT07046065
Title: Algorithm-assisted Subjective Refraction Program Dedicated to Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: WS10374; CIV-25-03-051757 (Other: INFARMED (Portugal))
Record Dates: First submitted 2025-06-12; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Refractive Assessment; Refractive Disorders; Hyperopia and Myopia; Astigmatism; Refractive Error Correction; Children
Keywords: cycloplegic refraction; non-cycloplegic refraction; subjective refraction
MeSH Terms: conditions — Refractive Errors; Hyperopia; Myopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Validation of the Kids Refraction softwares vA and vB performed with Vision-R™ phoropter (Active Comparator): Measurement of the non-cycloplegic refraction with Vision-R™ phoropter and comparison with the conventional refraction measurement method. Measurement of the cycloplegic refraction with Vision-R™ phoropter and comparison with non-cycloplegic refraction with Vision-R™ phoropter.
  Interventions: Device: Non-cycloplegic Objective refraction; Device: Non-cycloplegic conventional subjective refraction; Device: Non-cycloplegic subjective refraction (Kids refraction software vA with Vision-R™); Device: Non-cycloplegic subjective refraction (Kids refraction software vB with Vision-R™); Device: Cycloplegic subjective refraction (Kids refraction software vA with Vision-R™); Device: Cycloplegic Objective refraction; Device: Non-cycloplegic Retinoscopy; Device: Cycloplegic retinoscopy
- Validation of the Kids Refraction softwares vA and vB performed with Vision-S™ phoropter (Active Comparator): Measurement of the non-cycloplegic refraction with Vision-S™ phoropter and comparison with the conventional refraction measurement method. Measurement of the cycloplegic refraction with Vision-S™ phoropter and comparison with non-cycloplegic refraction with Vision-S™ phoropter.
  Interventions: Device: Non-cycloplegic Objective refraction; Device: Non-cycloplegic conventional subjective refraction; Device: Non-cycloplegic subjective refraction (Kids refraction software vA with Vision-S™); Device: Non-cycloplegic subjective refraction (Kids refraction software vB with Vision-S™); Device: Cycloplegic subjective refraction (Kids refraction software vA with Vision-S™); Device: Cycloplegic Objective refraction; Device: Non-cycloplegic Retinoscopy; Device: Cycloplegic retinoscopy

INTERVENTIONS:
Device: Non-cycloplegic Objective refraction — Objective refraction will be measured using an auto-kerato-refractometer/aberrometer without cyclopegia
Device: Non-cycloplegic conventional subjective refraction — Performed with Vision-R™
Device: Non-cycloplegic subjective refraction (Kids refraction software vA with Vision-R™) — Performed with Vision-R™
  Arms: Validation of the Kids Refraction softwares vA and vB performed with Vision-R™ phoropter
Device: Non-cycloplegic subjective refraction (Kids refraction software vA with Vision-S™) — Performed with Vision-S™
  Arms: Validation of the Kids Refraction softwares vA and vB performed with Vision-S™ phoropter
Device: Non-cycloplegic subjective refraction (Kids refraction software vB with Vision-R™) — Performed with Vision-R™
  Arms: Validation of the Kids Refraction softwares vA and vB performed with Vision-R™ phoropter
Device: Non-cycloplegic subjective refraction (Kids refraction software vB with Vision-S™) — Performed with Vision-S™
  Arms: Validation of the Kids Refraction softwares vA and vB performed with Vision-S™ phoropter
Device: Cycloplegic subjective refraction (Kids refraction software vA with Vision-R™) — Performed with Vision-R™
  Arms: Validation of the Kids Refraction softwares vA and vB performed with Vision-R™ phoropter
Device: Cycloplegic subjective refraction (Kids refraction software vA with Vision-S™) — Performed with Vision-S™
  Arms: Validation of the Kids Refraction softwares vA and vB performed with Vision-S™ phoropter
Device: Cycloplegic Objective refraction — Objective refraction will be measured using an auto-kerato-refractometer/aberrometer with cyclopegia
Device: Non-cycloplegic Retinoscopy — Performed with a retinoscope without cycloplegia
Device: Cycloplegic retinoscopy — Performed with a retinoscope with cycloplegia

SUMMARY:
Current refraction assessment in children is dependent on the Eye Care Specialist and lacks standardization. Essilor has developed new algorithm assisted subjective refraction software dedicated to children of 6-12 years old and suitable for use with Vision-S™ and Vision-R™ phoropters, in addition to existing software.

Two different versions of the software have been developed: the first incorporating only the steps needed to perform an entire subjective refraction process (vA), and the second, identical to the first but incorporating additional steps useful for managing the child's attention and cooperation (vB).

The software performance in terms of subjective refraction results will be compared to a conventional subjective refraction method performed with the Vision-R™700 phoropter in manual mode.

DETAILED DESCRIPTION:
The goal of the investigation is to evaluate the accuracy of the Kids refraction software results performed with the phoropters Vision-R™700 and Vision-S™700 compared to the conventional subjective refraction method results performed with Vision-R™700. Phase A of the investigation will focus on the validation of the first version (Kids refraction software vA), and phase B will involve the second version (Kids refraction software vB).

There are two phases in the investigation:

Phase A:

To evaluate the agreement of the subjective refraction results (Sphere, Cylinder, Axis, VA) between the Kids Refraction software vA (randomization between Vision-R or Vision-S devices) results and a conventional subjective refraction (performed with Vision-R), in a non-cycloplegic condition.

Phase B:

To evaluate the agreement of the subjective refraction results (Sphere, Cylinder, Axis, VA) between the Kids Refraction software vB with additional attention and cooperation stages (randomization between Vision-R or Vision-S devices) results and a conventional subjective refraction (performed with Vision-R), in a non-cycloplegic condition.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 and 12 years
2. Subject able to recognize and name the letters of the Latin alphabet
3. Pupillary distance (PD) not less than 49mm
4. Distance refractive error for spherical equivalence (SE) within the range of [-6.00 to +6.00 D] maximum of the two absolute values RE and LE; Cyl ≤ 3.00 D
5. Monocular Visual acuity ≥ +0.30 LogMAR (0.5 Decimal VA) in each eye at distance
6. Visual acuity difference < 0.20 logMAR between right and left eyes at distance

Exclusion Criteria:

1. Vulnerability of the subject
2. Amblyopia
3. Strabismus
4. Any current or evolving pathology manifested in the eye or the appendages which might have an influence on vision, or interfere with refractive state
5. Any previous ocular surgery, which might have an influence on vision or interfere with study assessments (e.g. iridectomy, refractive surgery…)
6. Any ocular or systemic condition known to affect refractive status (e.g., keratoconus, diabetes, Down's syndrome, etc.)
7. Any neurological or speech disorders that might interfere with the ability to understand and answer questions or communicate with the ECP
8. Any untreated and/or uncontrolled systemic condition which might have an influence on vision or interfere with study assessments
9. Current use of ocular or systemic medications, which, in the Investigator's opinion, may significantly affect pupil size, accommodation or refractive state
10. History of myopia control intervention that may affect refractive assessment (e.g., atropine, orthokeratology, rigid gas permeable lenses (RGP) etc.) except myopia control spectacles
11. Contraindications of cycloplegia (e.g. high Intra-ocular pressure - more than 22mmHg in either eye, narrow anterior angle, history of allergy to cycloplegic agents or seizures, etc)
12. Aphakic or pseudoaphakic (intraocular lens),
13. Prismatic prescription in either Right or Left eye (horizontal or vertical). -

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 166 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective Sphere (with Kids refraction software vA, with Vision-R™ and with Vision-S™) | Day 1
  The term "sphere" means that the correction for myopia or hyperopia is spherical, equal in all meridians of the eye. This indicates the amount of lens power, measured in diopters (D), prescribed to correct myopia or hyperopia.
Subjective Cylinder (with Kids refraction software vA, with Vision-R™ and with Vision-S™) | Day 1
  Indicates the amount of lens power for astigmatism, measured in diopters (D) and represents the difference in the greatest and weakest powers of the eye, usually separated by 90 degrees.
Subjective Axis (with Kids refraction software vA, with Vision-R™ and with Vision-S™) | Day 1
  Indicates the orientation of the Cylinder, measured in degrees (°)
Subjective Sphere (with Kids refraction software vB, with Vision-R™ and with Vision-S™) | Six months after Day 1
  The term "sphere" means that the correction for myopia or hyperopia is spherical, equal in all meridians of the eye. This indicates the amount of lens power, measured in diopters (D), prescribed to correct myopia or hyperopia.
Subjective Cylinder (with Kids refraction software vB, with Vision-R™ and with Vision-S™) | Six months after Day 1
  Indicates the amount of lens power for astigmatism, measured in diopters (D) and represents the difference in the greatest and weakest powers of the eye, usually separated by 90 degrees.
Subjective Axis (with Kids refraction software vB, with Vision-R™ and with Vision-S™) | Six months after Day 1
  Indicates the orientation of the Cylinder, measured in degrees (°)
Subjective Sphere (with conventional method with Vision-R™) | Day 1
  The term "sphere" means that the correction for myopia or hyperopia is spherical, equal in all meridians of the eye. This indicates the amount of lens power, measured in diopters (D), prescribed to correct myopia or hyperopia.
Subjective Cylinder (with conventional method, with Vision-R™) | Day 1
  Indicates the amount of lens power for astigmatism, measured in diopters (D) and represents the difference in the greatest and weakest powers of the eye, usually separated by 90 degrees.
Subjective Axis (with conventional method, with Vision-R™) | Day 1
  Indicates the orientation of the Cylinder, measured in degrees (°)
Visual acuity (with Kids refraction software vA, with Vision-R™ and with Vision-S™) | From enrollment (Day 1) to the end of the study at 7,5 months
  Corrected visual acuity measure with Kids refraction software vA results
Visual acuity (with Kids refraction software vB, with Vision-R™ and with Vision-S™) | From enrollment (Day 1) to the end of the study at 7,5 months
  Corrected visual acuity measure with Kids refraction software vB results
Visual acuity (with Conventionnal refraction method, with Vision-R™) | From enrollment (Day 1) to the end of the study at 7,5 months
  Corrected visual acuity measure with Conventionnal refraction method results

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel González- Meijome, PhD, Principal Investigator — Clinical & Experimental Optometry Research Lab Department of Physics (Optometry) - School of Science University of Minho, 4710-057 Gualtar - Braga (Portugal)
Locations (1):
- Centro de Investigação, Inovação e Ensino Superior (CIIES) de Famalicão, Vila Nova de Famalicão, Portugal

IPD SHARING:
Plan to Share IPD: No
There is no need to share individual anonymized data.